CLINICAL TRIAL: NCT03573869
Title: Effect of Cryoballoon Pulmonary Vein Isolation on Atrial Fibrillation Burden and Clinical Endpoints in Patients With Heart Failure With Impaired Left Ventricular Systolic Function
Brief Title: Atrial FIbrillation Treatment With Cryoballoon in Heart failurE (AFICHE)
Acronym: AFICHE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: G.Gennimatas General Hospital (Other)
Responsible Party: Principal Investigator, Spyridon Deftereos, Professor of Cardiology, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 39052/21-12-17
Record Dates: First submitted 2018-06-08; First posted 2018-06-29 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Atrial Fibrillation; Heart Failure, Systolic
MeSH Terms: conditions — Atrial Fibrillation; Heart Failure, Systolic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoballoon ablation (Experimental): A 28-mm cryoballoon (Arctic Front Advance™ Cardiac CryoAblation Catheter, Medtronic, Minneapolis, MN) will be employed. The cryoballoon catheter will be introduced into the left atrium, following a single transeptal puncture, through a 12F FlexCath steerable sheath (Medtronic), constantly flushed with heparinized saline. A circular mapping catheter (Achieve, Medtronic) will be advanced through the cryoballoon to the PV orifice and positioned as proximally as possible inside the vessel to record the PV potentials at baseline and monitor the isolation procedure in real time.
  Interventions: Procedure: Cryoballoon ablation
- Standard treatment (No Intervention): Standard treatment, including at least one rhythm control medication, on top of optimized rate control and HF treatment

INTERVENTIONS:
Procedure: Cryoballoon ablation — Left atrial ablation using cryoballoon to achieve pulmonary vein isolation
  Arms: Cryoballoon ablation

SUMMARY:
In this study 404 patients with heart failure and an ejection fraction of 0.40 or less, with paroxysmal atrial fibrillation, will be randomly assigned to standard treatment or standard treatment plus a session of cryoballoon ablation (left atrial balloon cryoablation for pulmonary vein isolation). All patients with either have an ICD or CRT-D/P device implanted or an implantable electrocardiographic monitoring device. The primary study endpoint will be the time to AF burden exceeding 1% over any 30-day period (calculated as the ratio of time spent in AF over total time).16 This AF burden corresponds to 7.2 hours per month.

A powered secondary endpoint will be the time to the composite of all-cause mortality and unplanned hospitalization for heart failure.

ELIGIBILITY:
Inclusion criteria:

* A minimum of at least two separate AF episodes recorded within the last 12 months, either on 12-lead rest ECG or on ambulatory ECG recordings (at least 5 minutes of AF on Holter recordings will be required),
* LVEF <40% on sinus rhythm,
* symptoms consistent with heart failure (New York Heart Association II or higher) despite rate control treatment,
* age >21 years old.

Exclusion criteria:

* previous left atrial ablation,
* left atrial diameter >28 mm/m2 BSA on TTE (parasternal long axis view),
* strong clinical suspicion that reduced LVEF is primarily due to tachycardiomyopathy,
* pre-existing device (ICD or CRT) without AF detection algorithms and/or (for CRT devices) diagnostics of effective biventricular pacing,
* known primary electrical heart disease (e.g. Brugada syndrome),
* presence of thrombus in a heart chamber,
* presence of prosthetic valve at any position,
* moderate/severe valvular heart disease,
* active infectious disease or malignancy,
* moderate or severe hepatic impairment (Child-Pugh class B or C),
* severe renal failure (estimated glomerular filtration rate <20 ml/min/1.73 m2),
* inability or unwillingness to adhere to standard treatment or to provide consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Time to exceed AG burden cut-off of 1% | Up to 2 years
  The time to AF burden exceeding 1% over any 30-day period (calculated as the ratio of time spent in AF over total time)

SECONDARY OUTCOMES:
All-cause mortality or hospitalization for heart failure | Up to 2 years
  Time to the composite of all-cause mortality and unplanned hospitalization for heart failure

CONTACTS AND LOCATIONS:
Locations (1):
- Athens General Hospital "G. Gennimatas", Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided